CLINICAL TRIAL: NCT01876420
Title: The Medtronic CoreValve™ Evolut R™ CE Mark Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT10093773DOC
Record Dates: First submitted 2013-06-05; First posted 2013-06-12 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The CoreValve™ Evolut R TAV™ system (Experimental): CoreValve™ Evolut R™ System which consists of the Evolut R™ Transcatheter Aortic Valve (26 & 29 mm sizes), EnVeo R™ Delivery Catheter System with Enveo InLine™ Sheath, and EnVeo R™ Loading System
  Interventions: Device: The CoreValve™ Evolut R TAV™ system

INTERVENTIONS:
Device: The CoreValve™ Evolut R TAV™ system — CoreValve™ Evolut R™ System which consists of the Evolut R™ Transcatheter Aortic Valve (26 & 29 mm sizes), EnVeo R™ Delivery Catheter System with Enveo InLine™ Sheath, and EnVeo R™ Loading System
  Other Names: CoreValve™ EvolutR™ Transcatheter Ao Valve; EnveoR™ Delivery Catheter System w/ Enveo InLine™ Sheath; EnVeoR™ Loding System

SUMMARY:
To assess the safety and clinical performance of the CoreValve™ Evolut R™ System.

DETAILED DESCRIPTION:
The study objectives are to assess the safety and clinical performance of the CoreValve™ Evolut R™ System in patients with severe symptomatic aortic stenosis who are considered at high through extreme risk for surgical aortic valve replacement. These objectives will be accomplished by a prospective clinical study involving up to 60 implanted subjects among up to six study centers.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis, defined as aortic valve area of < 1.0 cm2 (or aortic valve area index of < 0.6 cm2/m2) by the continuity equation, AND mean gradient > 40 mmHg or maximal aortic valve velocity > 4.0 m/sec by resting echocardiogram.
2. Estimated 30 day mortality risk of > 15% by study center Heart Team assessment,33 OR at least two cardiovascular surgeons from the study center deny surgery because of prohibitive operative risk, estimated to be a combined >50% risk of irreversible mortality or morbidity.
3. Symptoms of aortic stenosis, and NYHA Functional Class II or greater.
4. The subject meets the legal minimum age to provide informed consent based on local regulatory requirements, and has provided written informed consent as approved by the EC/IRB of the respective clinical site.
5. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

   Exclusion Criteria:

   Clinical exclusion criteria:
6. Subject has been offered SAVR but has declined.
7. Any condition considered a contraindication for placement of a bioprosthetic valve (e.g. subject is indicated for mechanical prosthetic valve).
8. Known hypersensitivity or contraindication to Nitinol.
9. Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
10. Untreated clinically significant coronary artery disease requiring revascularization.
11. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% by echocardiography, contrast ventriculography, or radionuclide ventriculography.
12. End stage renal disease requiring chronic dialysis of creatinine clearance < 20 cc/min.
13. Ongoing sepsis, including active endocarditis.
14. Any condition considered a contraindication to extracorporeal assistance.
15. Any percutaneous coronary or peripheral interventional procedure with a bare metal stent performed within 30 days prior to Heart Team assessment, or within six months prior to Heart Team assessment for procedures with a drug eluting stents.
16. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within eight weeks of Heart Team Assessment .
17. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
18. Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
19. Gastrointestinal (GI) bleeding that would preclude anticoagulation.
20. Subject refuses a blood transfusion.
21. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
22. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions.
23. Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol required follow-ups exams.
24. Currently participating in an investigational drug or another device study (excluding registries).
25. Evidence of an acute myocardial infarction ≤30 days before the index procedure.
26. Need for emergency surgery for any reason.
27. Liver failure (Child-C).
28. Subject is pregnant or breast feeding.

    Anatomical exclusion criteria:
29. Pre-existing prosthetic heart valve in any position.
30. Mixed aortic valve disease (aortic stenosis with moderate or severe aortic regurgitation).
31. Severe mitral regurgitation.
32. Severe tricuspid regurgitation.
33. Moderate or severe mitral stenosis.
34. Hypertrophic obstructive cardiomyopathy.
35. Echocardiographic or Multi-Slice Computed Tomography (MSCT) evidence of intracardiac mass thrombus or vegetation.
36. Congenital bicuspid or unicuspid valve verified by echocardiography.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vang, PhD, Study Director — Director Clinical Research Structural Heart
Locations (6):
- Australia (2):
  - Epworth Hospital, Melbourne, Victoria
  - Monash Medical Center, Melbourne, Victoria
- Waikato Hospital, Hamilton, New Zealand
- United Kingdom (3):
  - Royal Victoria Hospital, Belfast
  - Leeds General Infirmary, Leeds
  - St. George's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manoharan G, Walton AS, Brecker SJ, Pasupati S, Blackman DJ, Qiao H, Meredith IT. Treatment of Symptomatic Severe Aortic Stenosis With a Novel Resheathable Supra-Annular Self-Expanding Transcatheter Aortic Valve System. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1359-1367. doi: 10.1016/j.jcin.2015.05.015. PMID 26315740

RESULTS

PARTICIPANT FLOW:
Groups:
- All Implanted Subjects: Sixty subjects were implanted with the Evolut R valve from six centers in Australia, the United Kingdom, and New Zealand.
Period: Overall Study
Arm/Group | All Implanted Subjects
Started | 60
Completed | 59
Not Completed | 1
Not completed — Missed 30 day visit | 1

BASELINE CHARACTERISTICS:
Population: All implanted subjects
Arm/Group | The CoreValve™ Evolut R TAV™ System
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 20
Region of Enrollment [Number; unit: participants]
  New Zealand | 6
  United Kingdom | 29
  Australia | 25
NYHA Class [Number; unit: participants] — NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA) Class I Subject with cardiac disease but without resulting limitations of physical activity. Class II Subjects with cardiac disease resulting in slight limitation of physical activity. Class III Subjects with cardiac disease resulting in marked limitation of physical activity. Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  participants
    NYHA I | 0
    NYHA II | 19
    NYHA III | 36
    NYHA IV | 5
STS Score [Mean (Standard Deviation); unit: percent of risk for cardiac surgery] — The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  percent of risk for cardiac surgery | 7.0 (3.7)
Logistic EuroScore [Mean (Standard Deviation); unit: percent risk for cardiac surgery] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk.
  percent risk for cardiac surgery | 20.5 (12.5)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.7 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate at 30 Days
Description: The All-cause mortality rate at 30 days per the VARC II recommendation of clinical endpoints for TAVI. More specifically:
  Cardiovascular mortality (Any of the following criteria)
  * Death due to proximate cardiac cause (e.g. myocardial infarction, cardiac tamponade, worsening heart failure)
  * Death caused by non-coronary vascular conditions such as neurological events, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease
  * All procedure-related deaths, including those related to a complication of the procedure or treatment for a complication of the procedure
  * All valve-related deaths including structural or non-structural valve dysfunction or other valve-related adverse events
  * Sudden or unwitnessed death
  * Death of unknown cause Non-cardiovascular mortality
  * Any death in which the primary cause of death is clearly related to another condition (e.g. trauma, cancer, suicide)
Time Frame: 30 days
Population: All implanted subjects at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
percentage of participants | 0.0

2. Primary Outcome: Stroke Rate (Disabling and Non-disabling) at 30 Days
Description: The Stroke rate (disabling and non-disabling) at 30 days per the VARC II definitions. Stroke is defined as an acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of haemorrhage or infarction. Stroke may be classified as ischaemic or haemorrhagic with appropriate subdefinitions. Ischaemic stroke is defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue. Haemorrhagic stroke is defined as an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid haemorrhage. A stroke may be classified as 'undetermined' if there is insufficient information to allow the categorization as ischaemic or haemorrhagic.
Time Frame: 30 days
Population: All implanted subjects at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
percentage of participants | 0.0

3. Primary Outcome: Device Success Rate at 24 Hours to Seven Days
Description: 1. Device success rate at 24 hours to seven days, defined as:
     * Absence of procedural mortality, AND
     * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
     * Intended performance of the prosthetic heart valve, defined as the absence of patient-prosthesis-mismatch and mean aortic valve gradient less than 20 mmHg (or peak velocity < 3 m/sec), AND absence of moderate or severe prosthetic valve regurgitation.
  2. The percentage of subjects with no more than mild aortic regurgitation at early post procedure echocardiogram (24 hours through seven days).
Time Frame: 24 hours to seven days
Population: All implanted subjects at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
percentage of participants
  Overall Device Success | 78.6
  Absence of Procedural Mortality | 100.0
  Correct Positioning of Single Valve | 98.3
  Intended Performance of Prosthetic Heart Valve | 80.0
  Absence of Patient Prosthesis Mismatch | 83.6
  Mean Gradient < 20mmHg or Peak Velocity < 3m/sec | 98.3
  Absence of Mod. or Severe Prosthetic Regurgitation | 93.3

4. Secondary Outcome: VARC II Combined Safety Endpoint at 30 Days
Description: The VARC II Combined Safety Endpoint at 30 days includes the following components: All-Cause Mortality, All Stroke, Life Threatening or Disabling Bleeding, Acute Kidney Injury: Stage 2 or 3, Coronary Artery Obstruction, Major Vascular Complication, and Valve-Related Dysfunction Requiring Repeat Procedure.
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
percentage probability | 13.3

5. Secondary Outcome: Event Rates of the Individual Components of the VARC II Composite Safety Endpoint at 30 Days
Description: The Individual components of the VARC II composite safety endpoint at 30 days per the Kaplan Meier Event Rate (%).
Time Frame: 30 days
Population: The number of subjects analyzed at 30 days.
Measure: Number; unit: percentage of probability
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
percentage of probability
  Combined Safety Endpoint | 13.3
  All Cause Mortality | 0.0
  All Stroke | 0.0
  Life Threatening or Disabling Bleeding | 5.0
  Acute Kidney Injury: Stage 2 or 3 | 1.7
  Coronary Artery Obstruction | 0.0
  Major Vascular Complication | 8.3
  Valve-Related Dysfunct. Requiring Repeat Procedure | 0.0

6. Secondary Outcome: Hemodynamic Performance Metrics at 30 Days by Doppler Echocardiography - Mean Gradient
Description: The hemodynamic performance will be measured by the Mean Prosthetic Valve Gradient for 59 subjects, measured with the Doppler echocardiography.
Time Frame: 30 days
Population: All implanted subjects who had echos at the 30 day visit, which were 58 subjects, only 57 of the echos were able to measure the Mean Gradient for those subjects.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 57
mmHg | 8.1 (3.3)

7. Secondary Outcome: Hemodynamic Performance Metrics at 30 Days by Doppler Echocardiography - • Effective Orifice Area (EOA)
Description: Effective orifice area
Time Frame: 30 days
Population: All implanted subjects who had echos at the 30 day visit, which were 58 subjects, only 54 of the echos were able to measure the EOA for those subjects.
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 54
cm² | 1.9 (0.5)

8. Secondary Outcome: Hemodynamic Performance Metrics at 30 Days by Doppler Echocardiography - Total Aortic Regurgitation (Transvalvular & Paravalvular)
Description: Degree of Total prosthetic valve regurgitation (transvalvular & paravalvular)
Time Frame: 30 days
Population: All implanted subjects who had echos at the 30 day visit, which were 58 subjects, and 58 of the echos were able to measure the Total Aortic Regurgitation for those subjects.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 58
percentage of participants
  None | 8.6
  Trace | 22.4
  Mild | 63.8
  Moderate | 5.2
  Severe | 0.0

9. Secondary Outcome: Resheath or Recapture Success Rate (When Attempted), Where Successful Recapture is Defined as Evolut R™ TAV (Including the Frame) is Fully Resheathed Into the Capsule of the Delivery Catheter, as Verified by Fluoroscopy.
Description: Resheath or Recapture success rate (when attempted), where successful recapture is defined as Evolut R™ TAV (including the frame) is fully resheathed into the capsule of the delivery catheter, as verified by fluoroscopy. Resheathing or recapturing of the TAV was attempted on 15 subjects.
Time Frame: Day 1
Population: Subjects who had either a resheath or recapture attempt at implant and the success rate for each resheathing, or recapturing attempts of the valve at the implant.
Measure: Number; unit: percentage of successful attempts
Units Other Than Participants: Research recapture attempts
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 15
Number analyzed (Research recapture attempts) | 22
percentage of successful attempts
  Success rate for Resheath or Recapture | 100.0
  Success rate for Resheath | 100.0
  Success rate for Recapture | 100.0

ADVERSE EVENTS:
Time Frame: Up to 30 days.
Description: All SAE should be reported as soon as possible, not later than within ten days of knowledge of the event. All other adverse events should be reported as soon as possible, not later than within three weeks.
Groups:
- All Attempted Implanted Subjects: Sixty subjects were implanted with the Evolut R valve from six centers in Australia, the United Kingdom, and New Zealand.
Arm/Group | All Attempted Implanted Subjects
Serious Adverse Events (participants affected / at risk) | 40/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Attempted Implanted Subjects (N=60)
Anemia (Blood and lymphatic system disorders) | 3
Blood disorder (Blood and lymphatic system disorders) | 1
Cardiac Conduction Disorder (Cardiac disorders) | 8
Supraventricular arrythmia (Cardiac disorders) | 1
Pulmonary edema (Cardiac disorders) | 1
Ischemic Coronary Artery Disorder (Cardiac disorders) | 1
Decreased BP (Cardiac disorders) | 1
Gastrointestianl Ulcers and Perforation, Site Unspecified (Gastrointestinal disorders) | 2
General Signs and Symptoms Nec (General disorders) | 1
Infections (Infections and infestations) | 4
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 1
Complications (Injury, poisoning and procedural complications) | 12
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Renal Failure and Impairment (Renal and urinary disorders) | 1
Upper Respiratory Tract Signs and Symptoms (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Ascribed to Specific Agent (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Attempted Implanted Subjects (N=60)
Anaemias Nec (Blood and lymphatic system disorders) | 5
Thrombocytopenias (Blood and lymphatic system disorders) | 2
Cardiac Conduction Disorders (Cardiac disorders) | 29
Cardiac Disorders Nec (Cardiac disorders) | 12
Heart Failure Nec (Cardiac disorders) | 3
Ischemic Coronary Artery Disorders (Cardiac disorders) | 2
Rate and Rhythm Disorders (Cardiac disorders) | 4
Supraventricular Arrythmias (Cardiac disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal Atonic And Hypomobility (Gastrointestinal disorders) | 5
Nausea and Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal Atonic And HypomobilitySigns and Symptoms Nec (Gastrointestinal disorders) | 2
Febrile Disorders (General disorders) | 1
Inflammations (General disorders) | 1
Complication Associated with Device Nec (General disorders) | 1
Infections Nec (Infections and infestations) | 6
Urinary Tract Infections (Infections and infestations) | 8
Non-site specific Injuries Nec (Injury, poisoning and procedural complications) | 6
Non-site specific Procedural Complications (Injury, poisoning and procedural complications) | 8
General Nutrition Disorders (Metabolism and nutrition disorders) | 17
Headach Nec (Nervous system disorders) | 2
Neurological Signs And Symptoms Nec (Nervous system disorders) | 1
Depressive Disorders (Psychiatric disorders) | 1
Mental Disorder (Psychiatric disorders) | 4
Renal Failure and Impairment (Renal and urinary disorders) | 2
Urinary Abnormalities (Renal and urinary disorders) | 2
Vulvovaginal Disorder Nec (Reproductive system and breast disorders) | 1
Coughing And Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax And Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 4
Dermatitis And Eczema (Skin and subcutaneous tissue disorders) | 1
Subcutaneous Tissue Ulcerations (Skin and subcutaneous tissue disorders) | 3
Skin injuries And Mechanical Dermatoses (Skin and subcutaneous tissue disorders) | 4
Vascular Hypotensive Disorders (Vascular disorders) | 4
Aortic Valvular Disorders (Cardiac disorders) | 2
Ventricular Arrythmias (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No